CLINICAL TRIAL: NCT06585917
Title: A Multicenter Study Comparing the Efficacy and Safety of 6F and 7F Thin-Walled Sheaths Via Distal Radial Artery Access for Coronary Intervention
Brief Title: Comparison of 6F and 7F Sheaths for Coronary Intervention Via Distal Radial Artery Access
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-2377
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-09

CONDITIONS: PCI; Coronary Arterial Disease (CAD)
Keywords: Distal Radial Artery Access; Coronary Intervention; 7F Sheath; 6F Sheath; Radial Artery Occlusion; Non-Inferiority Trial
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: This study uses a Parallel Assignment model, where participants are randomly assigned to one of two groups: the 7F sheath intervention group or the 6F sheath control group. Each group will receive a different size sheath for coronary intervention via distal radial artery access. The study is designed to compare the outcomes between these two groups, with no crossover between groups during the trial. This model allows for a direct comparison of the efficacy and safety between the two sheath sizes under similar clinical conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 7F Sheath Intervention Group (Experimental): Participants in this arm will undergo coronary intervention using a 7F thin-walled sheath via distal radial artery access. This group will be used to assess the efficacy and safety of the 7F sheath compared to the 6F sheath.
  Interventions: Device: 7F Thin-Walled Sheath
- 6F Sheath Control Group (Active Comparator): Participants in this arm will undergo coronary intervention using a 6F thin-walled sheath via distal radial artery access. This group will serve as the control to compare the outcomes against those of the 7F sheath group.
  Interventions: Device: 6F Thin-Walled Sheath

INTERVENTIONS:
Device: 7F Thin-Walled Sheath — The 7F Thin-Walled Sheath is used during coronary intervention procedures via distal radial artery access. This device has a smaller outer diameter compared to traditional 7F sheaths, designed to reduce the risk of vascular complications while allowing for the performance of complex coronary interventions.
  Arms: 7F Sheath Intervention Group
Device: 6F Thin-Walled Sheath — The 6F Thin-Walled Sheath is the standard device used in coronary intervention procedures via distal radial artery access. It is employed as a control in this study to compare its efficacy and safety against the 7F Thin-Walled Sheath.
  Arms: 6F Sheath Control Group

SUMMARY:
This is a multicenter, randomized controlled, prospective, non-inferiority, open-label study aiming to evaluate whether the efficacy and safety of using a 7F thin-walled sheath via distal radial artery (dTRA) access for coronary intervention (PCI) are non-inferior to the use of a 6F thin-walled sheath. The study population includes adult patients who are candidates for coronary intervention. The primary endpoint is the rate of radial artery and distal radial artery occlusion 24 hours post-procedure.

DETAILED DESCRIPTION:
This study is a multicenter, randomized controlled, prospective, non-inferiority, open-label clinical trial designed to compare the efficacy and safety of using 7F thin-walled sheaths versus 6F thin-walled sheaths for coronary intervention (PCI) via distal radial artery access (dTRA). The study will enroll adult patients with coronary artery disease who are scheduled to undergo PCI.

Participants will be randomized into two groups: the experimental group, which will receive PCI using a 7F sheath, and the control group, which will receive PCI using a 6F sheath. The primary endpoint is the rate of radial artery and distal radial artery occlusion 24 hours post-procedure, assessed by ultrasound. Secondary endpoints include the incidence of major adverse cardiovascular and cerebrovascular events during follow-up, cannulation success rate, PCI success rate, and the rate of radial artery occlusion at 30 days post-procedure, among others.

The study aims to determine whether the 7F sheath is non-inferior to the 6F sheath in terms of safety and efficacy for PCI through dTRA. The study will be conducted at multiple centers in China, with a planned enrollment of 574 participants, and it will span from Sep 2024 to January 2026. All procedures will adhere to the highest standards of clinical practice, and patient data will be managed with strict confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤80 years;
* Height ≤180 cm;
* Distal radial artery diameter ≥1.7 mm;
* Completed distal radial artery angiography and requires coronary intervention;
* Tolerates dual antiplatelet therapy and intraoperative anticoagulant therapy, with no history of related drug allergies;
* Patient consents to participate in the study.

Exclusion Criteria:

* Acute myocardial infarction requiring emergency PCI;
* Ultrasound-confirmed occlusion of the radial artery on the procedure side;
* Radial artery and distal radial artery anomalies (e.g., small caliber, tortuous, looped vessels) that make the dTRA approach unsuitable;
* Previous bilateral radial artery intervention or surgery;
* No coronary intervention performed after coronary angiography;
* Inability to undergo coronary angiography and intervention due to subjective or objective reasons;
* Coronary lesions requiring the use of a 7F guiding catheter;
* Coronary arteries not suitable for 7F guiding catheter;
* Severe liver or renal insufficiency, unresolved bleeding disorders, or other serious conditions with an expected survival of less than 1 year;
* Currently breastfeeding or known pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Radial Artery Occlusion Rate 24 Hours Post-Procedure | 24 hours post-procedure
  The primary outcome is the rate of radial artery and distal radial artery occlusion 24 hours after the procedure. Occlusion will be determined by the absence of blood flow spectrum in the radial artery as assessed by ultrasound.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | Up to 30 days post-procedure
  The incidence of major adverse cardiovascular and cerebrovascular events during the follow-up period, including all-cause mortality, cardiovascular mortality, new-onset myocardial infarction, and new-onset stroke.
Cannulation Success Rate | During the procedure
  The success rate of sheath insertion and placement in the radial artery during the coronary intervention procedure.
PCI Success Rate | During the procedure
  The success rate of the percutaneous coronary intervention (PCI) procedure, defined by the successful completion of the intended intervention with appropriate device placement and without the need for conversion to an alternative access site.
Radial Artery Occlusion Rate 30 Days Post-Procedure | 30 days post-procedure
  The rate of radial artery and distal radial artery occlusion 30 days after the procedure, assessed by ultrasound.
Major Bleeding Events | Up to 30 days post-procedure
  The incidence of major bleeding events, defined according to the Bleeding Academic Research Consortium (BARC) criteria (Type 3 or Type 5 bleeding).
Local Neurological Complications | Up to 30 days post-procedure
  The incidence of local neurological complications, including numbness, tingling, or motor deficits in the arm used for radial artery access.
Incidence and Severity of Forearm Hematoma | Up to 30 days post-procedure
  Forearm hematoma will be graded using the EASY (Early Discharge After Transradial Stenting of Coronary Arteries Study) hematoma scale. The scale ranges from Grade I to Grade V:
  Grade I: Hematoma <5 cm in diameter (non-significant) Grade II: Hematoma 5-10 cm in diameter (mild) Grade III: Hematoma >10 cm but distal to the elbow (moderate) Grade IV: Hematoma extending above the elbow (severe) Grade V: Hematoma associated with ischemic threat to the hand (compartment syndrome) Higher grades indicate worse outcomes.
Pain Scores | Up to 30 days post-procedure
  Patient-reported pain scores assessed using the Visual Analog Scale (VAS). The scale ranges from 0 (no pain) to 10 (worst pain), with higher scores indicating worse outcomes.
Daily Living Ability Scores | Up to 30 days post-procedure
  Daily living abilities assessed using the Barthel Index, which ranges from 0 (complete dependence) to 100 (complete independence), with higher scores indicating better outcomes.
Length of Hospital Stay | From the time of admission for the procedure until the date of discharge, assessed up to 30 days post-procedure
  The total length of hospital stay, measured in days, starting from the date of admission for the coronary intervention procedure until the date of discharge, with a maximum assessment period of up to 30 days post-procedure.
Unplanned Additional Interventions During Hospitalization | From the time of procedure until discharge, assessed up to 30 days post-procedure
  The incidence of unplanned additional interventions required during the initial hospitalization, including but not limited to additional PCI, vascular repair, or treatment of complications. The events will be assessed from the time of the procedure until the patient is discharged, with a maximum assessment period of up to 30 days post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Lijian Gao, PhD. MD., Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences
Locations (1):
- Fuwai Hospital, CAMS & PUMC, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The decision not to share individual participant data (IPD) is based on concerns related to patient confidentiality and data privacy. While all data collected in this study will be securely stored and managed, the nature of the data involves sensitive health information that could potentially identify participants. Furthermore, the current study does not have the necessary infrastructure or resources in place to manage the secure and controlled distribution of IPD to external researchers. Therefore, to protect participant privacy and adhere to ethical standards, we have decided not to share IPD for this trial.

REFERENCES:
- [Derived] Liu M, Du Y, Cui C, Li C, Yu W, Wang H, Song Y, Gao Z, Song L, Zhai J, Yang Y, Yang W, Wu Y, Liu D, Guo J, Heisha N, Liu H, Zhao Y, Zhang F, Tang Y, Zhao Y, Yu M, Zhang B, Yang J, Li R, Li H, Xiong X, Guo X, Li H, Song Y, Duan F, Gao L. Distal Radial Artery Access With 6F and 7F Thin-Walled Sheaths for Coronary Intervention: A Multicentre, Randomized, DRAWS Trial Protocol. Can J Cardiol. 2025 Dec;41(12):2420-2428. doi: 10.1016/j.cjca.2025.09.002. Epub 2025 Sep 13. PMID 40953816